CLINICAL TRIAL: NCT04678050
Title: Dexmedetomidine Compared to Ketofol for Sedation in Paediatrics Undergoing Dental Procedures: a Comparative Study
Brief Title: Dexmedetomidine Compared to Ketofol for Sedation in Paediatrics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, MD, Lecturer of Anaesthesia and intensive care, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB 000-6379
Record Dates: First submitted 2020-12-03; First posted 2020-12-21 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Vital Signs
MeSH Terms: interventions — Ketamine; Propofol; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: The study participants will be allocated into two equal groups. Subjects in group I will receive ketofol solution (ketamine/propofol mixture, each mL contains 5 mg of ketamine plus 10 mg of propofol). A loading dose of 0.125 mL/kg will be administered intravenously (IV) over 10 min, followed by maintenance infusion at a rate of 0.05-0.125 mL/kg/h. Subjects in group II will receive the Dex solution (4 µg/mL). A loading dose of 2 µg/kg will be administered IV over 10 min, followed by a maintenance infusion of 0.1-1 µg/kg/h. Non-invasive blood pressure (mean ABP) peripheral oxygen saturation, heart rate, and respiratory rate will be assessed at baseline, at 2 minutes, then at 5 minutes intervals till 60 minutes. Ramsay sedation and Aldrete's recovery rating scores were assessed before, during, and after the procedure.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pedo-dentist, the independent observer/data collector, and participants will be blind to the type of intervention. The study drugs will be prepared by an anesthesiologist who will not participate in the observation of the data. All the lines and syringes will be wrapped to mask colors of the sedative drugs, and the syringes will be label coded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group I received ketamine/propofol (ketofol) solution (Active Comparator): ketamine/propofol mixture, each mL contains 5 mg of ketamine plus 10 mg of propofol). A loading dose of 0.125 mL/kg will be administered intravenously (IV) over 10 min, followed by maintenance infusion at a rate of 0.05-0.125 mL/kg/h.
  Interventions: Drug: Ketamine/ propofol
- group II received the Dex solution (4 µg/mL (Active Comparator): A loading dose of 2 µg/kg will be administered IV over 10 min, followed by a maintenance infusion of 0.1-1 µg/kg/h.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Ketamine/ propofol — ketamine/propofol mixture, each mL contains 5 mg of ketamine plus 10 mg of propofol). A loading dose of 0.125 mL/kg will be administered intravenously (IV) over 10 min, followed by maintenance infusion at a rate of 0.05-0.125 mL/kg/h.
  Other Names: Ketofol
  Arms: group I received ketamine/propofol (ketofol) solution
Drug: Dexmedetomidine — Dex solution (4 µg/mL). A loading dose of 2 µg/kg will be administered IV over 10 min, followed by a maintenance infusion of 0.1-1 µg/kg/h
  Other Names: precedex
  Arms: group II received the Dex solution (4 µg/mL

SUMMARY:
Dental fear and anxiety remain common problems that should be managed by both the dentist and the anesthetist. The currently available evidence for safe and effective sedative drugs for children undergoing the dental procedure is scarce The aim of this study was to compare the safety and efficacy of intravenous ketofol versus dexmedetomidine (Dex) as premedications a sedative in anxious children undergoing dental pulp therapy

DETAILED DESCRIPTION:
This double-blind, parallel-group, randomized clinical study will recruiter anxious children who will undergo dental pulp therapy. The study participants will be allocated into two equal groups. Subjects in group I will receive ketofol solution (ketamine/propofol mixture, each mL contains 5 mg of ketamine plus 10 mg of propofol). A loading dose of 0.125 mL/kg will be administered intravenously (IV) over 10 min, followed by maintenance infusion at a rate of 0.05-0.125 mL/kg/h. Subjects in group II will receive the Dex solution (4 µg/mL). A loading dose of 2 µg/kg will be administered IV over 10 min, followed by a maintenance infusion of 0.1-1 µg/kg/h. Non-invasive blood pressure (mean ABP), peripheral oxygen saturation, heart rate, and respiratory rate will be assessed at baseline, at 2 minutes, then at 5 minutes intervals till 60 minutes. Ramsay sedation and Aldrete's recovery rating scores will be assessed before, during, and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* ASA-I children,
* aged 5-10 years-old,
* requiring dental pulp therapy

Exclusion Criteria:

* ASA class ≥ II;
* previous experience with GA or Conscious sedation (CS);
* dental treatment expected to exceed 45 minutes;
* history of allergy to local anesthetics, Dex, propofol, ketamine, eggs, or soya;
* respiratory tract infections

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
the Number of interruptions | through study completion, an average of 3 month
  the Number of interruptions that occurred during the procedure

SECONDARY OUTCOMES:
total dose of rescue drug | through study completion, an average of 3 month
  total dose of rescue propofol in mg

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Ismail, MD, Study Chair — Head of research ethics committee
Locations (1):
- Ain Shams University, Cairo, Abassia, Egypt

IPD SHARING:
Plan to Share IPD: No